CLINICAL TRIAL: NCT02945124
Title: The Effects of K-Tape on Walking Pattern, Muscle Activity, and Motor Performance in Children With and Without Developmental Coordination Disorder: a Randomized Controlled Trial
Brief Title: Taping for Children With and Without Movement Clumsiness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA1512037
Record Dates: First submitted 2016-09-10; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Developmental Coordination Disorder
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Normal children with K Tape (Experimental)
  Interventions: Other: K tape
- Normal children without K Tape (No Intervention)
- DCD with K Tape (Experimental)
  Interventions: Other: K tape
- DCD without K Tape (No Intervention)

INTERVENTIONS:
Other: K tape — Applying K tape to children to the lower limb muscles during motor activities.
  Arms: DCD with K Tape; Normal children with K Tape

SUMMARY:
To investigate the effects of K Tape on walking pattern, muscle activity and motor performance in children with and without developmental coordination disorder (DCD).

ELIGIBILITY:
Inclusion Criteria:

* Children with DCD and typically developing children will need to score <16 percentile and >25 percentile, respectively, on MABC-2
* Study in mainstream schools
* No intellectual disabilities

Exclusion Criteria:

* Subjects who are receiving regular treatments
* Demonstrate excessive disruptive behaviour
* Unable to follow instructions
* Any diagnosis of neurological, musculoskeletal or cognitive disorder that affects test performance

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in lower limb muscle activation as measured by electromyography | Day 1 and day 2 (ms)
  Post K Tape lower limb muscle activity - pre K Tape lower limb muscle activation

SECONDARY OUTCOMES:
Change in balance performance as measured by force plate | Day 1 and day 2
  Post K Tape balance performance - pre K Tape balance performance
Foot posture as assessed by clinical observation | Day 1 and Day 2
Body composition as assessed by DXA | Day 1 and Day 2
Change in walking pattern as assessed by a motion analysis system | Day 1 and day 2
  Post K Tape walking pattern - pre K Tape walking pattern

CONTACTS AND LOCATIONS:
Overall Officials: Siu Ming Fong, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Pokfulam, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fong SSM, Ng SSM, Guo X, Wang Y, Chung RCK, Stat G, Ki WY, Macfarlane DJ. Deficits in Lower Limb Muscle Reflex Contraction Latency and Peak Force Are Associated With Impairments in Postural Control and Gross Motor Skills of Children With Developmental Coordination Disorder: A Cross-Sectional Study. Medicine (Baltimore). 2015 Oct;94(41):e1785. doi: 10.1097/MD.0000000000001785. PMID 26469921